CLINICAL TRIAL: NCT06495021
Title: OMT and Respiratory Illness
Brief Title: How OMT Benefits Newly Diagnosed Patients With Respiratory Illness When Given Alongside Other Standard Care.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0453
Record Dates: First submitted 2024-07-03; First posted 2024-07-10 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Pneumonia; Sinusitis; Bronchitis; Respiratory Disease; Respiratory Tract Infections
Keywords: Osteopathic Manual Therapy; Respiratory Illness; OMT
MeSH Terms: conditions — Pneumonia; Sinusitis; Bronchitis; Respiration Disorders; Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into a control group and treatment group for their duration of the study upon informed consent. Control patients will not receive lymphatic pump OMT, while treatment patients will receive lymphatic pump therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients in the control group will receive normal standard care, including any prescriptions, follow-up instructions, etc., as given by the provider to help treat their condition.
- Treatment (Experimental): Patients will receive lymphatic pump OMT therapy in addition to other standard care (similar to the control patients, this would be a medication, follow-up instructions, etc.)
  Interventions: Procedure: Lymphatic Pump Osteopathic Manipulative Therapy

INTERVENTIONS:
Procedure: Lymphatic Pump Osteopathic Manipulative Therapy — OMT is a series of manual pressure and physical stimulation among various parts of the body to stimulate fluid movement and immune response in patients with various symptoms and disease. This may help with conditions such as edema, clearance of infections, facilitate healing and circulation, and bolster the immune response. Specifically, the lymphatic pump type of OMT targets the head, neck, thoracic region, lumbar and sacral regions, pelvis, arms, legs, and abdomen.
  Other Names: Lymphatic Pump OMT
  Arms: Treatment

SUMMARY:
This study is to see Osteopathic Manipulative Therapy, or OMT, can aid in treating patients being seen for respiratory illness and associated symptoms. The hypothesis is that the addition of OMT therapy, alongside other standard care (such as a medication), can help lessen patient symptoms sooner than just other treatment alone, and the duration of the condition will shorten as well.

DETAILED DESCRIPTION:
Respiratory illness is a common complaint seen routinely in primary care. Illness is a common cause of reduced productivity, general discomfort and missed time from work. Osteopathic manual therapy (OMT) and the lymphatic pump is used frequently among osteopathic physicians to treat patients with infections. Many osteopathic physicians have anecdotal reports of patient having reduced respiratory symptoms reported in follow up care from patients. OMT is a useful, low-cost treatment and can help reduce duration of illness symptoms, improve patients' comfort and accelerate their return to their productive lives.

There have been few studies on an outpatient level quantifying this improvement. Previous research in other models have showed benefits of OMT to help reduce illness. Studies in a rat model have shown reduced S. pneumonia bacterial load in the lung after lymphatic pump. Additional rat studies demonstrated improved benefit with lymphatic pump in addition to antibiotic treatment. In a dog model, lymphatic pump has been shown to increase cytokine flow to the thoracic duct. In humans, OMT has shown to improve secretory immunoglobulin A levels in stressed student population. In the hospital setting, OMT for patients with pneumonia has shown to decrease hospital length of stay 5. OMT has been a known useful additional treatment to pneumonia, however there are few prospective studies on treatment of pneumonia and respiratory illness in the outpatient setting.

This study is designed to support evidence that patients with a recent diagnosis of upper respiratory illness, sinusitis, bronchitis, or pneumonia who receive lymphatic pump OMT experience reduced severity and length of symptoms. After informed consent, patients of ages 65-100 years of age who are diagnosed with a respiratory illness will be randomized to either standard care without OMT, or standard care plus OMT. Patients will be provided an electronic survey to quantify symptoms of cough, congestion, and malaise on both the day of illness diagnosis followed by the same survey 5 days later. Survey results comparing day of diagnosis and 5 days later will be recorded in a secure database and analyzed with appropriate statistical testing. The goal of this study is to show how the lymphatic pump can reduce both severity and duration of symptoms related to respiratory illness.

ELIGIBILITY:
Inclusion Criteria:

* Patients being seen for respiratory illness symptoms at Geisinger 65-Forward Buckhorn, PA clinic for care.
* Patients age of 65-100
* New diagnosis of upper respiratory illness, sinusitis, bronchitis, or pneumonia during outpatient visit.

Exclusion Criteria:

* Patients that have a healing fracture, including the spine, pelvis, shoulder, ribs, vertebrae, or extremities.
* Patients actively receiving any type of cancer treatment
* Patients with active or previously diagnosed liver disease.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
To address the magnitude in which lymphatic pump OMT improves respiratory illness symptom severity and overall sickness duration when combined with standard care treatment. | Through study completion of up to one year.
  Survey given to patients will provide feedback to capture their symptom severity at the time of diagnosis and 5 days post-diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Moore, DO, Principal Investigator — Physician
Locations (1):
- Geisinger 65-Forward, Buckhorn, Bloomsburg, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is no direct intent to share individual participant data related to this study. However, per institute policy, records of data generated during this study will be de-identified and will be kept for at least 6 years within the institutes secured database and then destroyed. Prior to destruction, the data will have the OPTION of being used for other Geisinger institutional review board-approved research if appropriate.

REFERENCES:
- [Background] Creasy C, Schander A, Orlowski A, Hodge LM. Thoracic and abdominal lymphatic pump techniques inhibit the growth of S. pneumoniae bacteria in the lungs of rats. Lymphat Res Biol. 2013 Sep;11(3):183-6. doi: 10.1089/lrb.2013.0007. Epub 2013 Sep 11. PMID 24024572
- [Background] Hodge LM, Creasy C, Carter K, Orlowski A, Schander A, King HH. Lymphatic pump treatment as an adjunct to antibiotics for pneumonia in a rat model. J Am Osteopath Assoc. 2015 May;115(5):306-16. doi: 10.7556/jaoa.2015.061. PMID 25938525
- [Background] Knott EM, Tune JD, Stoll ST, Downey HF. Increased lymphatic flow in the thoracic duct during manipulative intervention. J Am Osteopath Assoc. 2005 Oct;105(10):447-56. PMID 16314677
- [Background] Saggio G, Docimo S, Pilc J, Norton J, Gilliar W. Impact of osteopathic manipulative treatment on secretory immunoglobulin a levels in a stressed population. J Am Osteopath Assoc. 2011 Mar;111(3):143-7. PMID 21464262
- [Background] Noll DR, Degenhardt BF, Fossum C, Hensel K. Clinical and research protocol for osteopathic manipulative treatment of elderly patients with pneumonia. J Am Osteopath Assoc. 2008 Sep;108(9):508-16. PMID 18806080
- [Background] Noll DR, Degenhardt BF, Johnson JC. Multicenter Osteopathic Pneumonia Study in the Elderly: Subgroup Analysis on Hospital Length of Stay, Ventilator-Dependent Respiratory Failure Rate, and In-hospital Mortality Rate. J Am Osteopath Assoc. 2016 Sep 1;116(9):574-87. doi: 10.7556/jaoa.2016.117. PMID 27571294
- [Background] Yao S, Hassani J, Gagne M, George G, Gilliar W. Osteopathic manipulative treatment as a useful adjunctive tool for pneumonia. J Vis Exp. 2014 May 6;(87):50687. doi: 10.3791/50687. PMID 24836893
- [Background] Noll DR. The short-term effect of a lymphatic pump protocol on blood cell counts in nursing home residents with limited mobility: a pilot study. J Am Osteopath Assoc. 2013 Jul;113(7):520-8. doi: 10.7556/jaoa.2013.003. PMID 23843375
- [Background] Becker AD. Osteopathic treatment of the common cold. 1937. J Am Osteopath Assoc. 2001 Aug;101(8):461-3. No abstract available. PMID 11534526